CLINICAL TRIAL: NCT05053399
Title: Evaluation of Clinical Outcomes in China for the TECNIS Symfony® Toric Intraocular Lens Model Series ZXT
Brief Title: Evaluation of the TECNIS Symfony® Toric Intraocular Lens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Surgical Vision, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PCOL-202-CHSF
Record Dates: First submitted 2021-09-16; First posted 2021-09-22 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Cataracts
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TECNIS Symfony Toric IOL (Experimental): Model Series ZXT
  Interventions: Device: Model Series ZXT

INTERVENTIONS:
Device: Model Series ZXT — Investigational intraocular lens replaces the natural lens removed during cataract surgery in both eyes.

SUMMARY:
This is a prospective, single-center, single-arm, open-label, clinical study of the investigational TECNIS Symfony® Toric IOL. The study will enroll up to 100 subjects from a single investigative site in China. The subjects will be followed for 12-months postoperatively.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients at least 18 years of age
2. Have a cataract in one or both eyes, with planned phacoemulsification with intraocular lens implantation
3. Have estimated postoperative visual acuity of at least 20/25 Snellen (0.8 decimal) in the eye to be implanted per surgeon estimate \
4. Regular corneal astigmatism and predicted postoperative residual astigmatism of less than 1.00 D after implantation with a toric intraocular in the study eye(s)
5. Availability, willingness and sufficient cognitive awareness to understand the purpose of the examination procedures and comply with postoperative visits that are required by the study protocol
6. Voluntary participation indicated by the study informed consent form (ICF) signed by the patient or legal guardian.

Exclusion Criteria:

1. Concurrent participation or participation in any other clinical study within 30 days prior to the preoperative visit
2. Ocular disease (other than cataract) that may significantly affect postoperative vision, such as visually significant keratopathy, macular lesions, diabetic retinopathy, chronic or severe uveitis, etc.
3. Prior corneal refractive (LASIK, LASEK, RK, PRK, etc.) or intraocular surgery, including prophylactic peripheral iridotomies and peripheral laser retinal repairs
4. Irregular corneal astigmatism
5. Inability to achieve keratometric stability for contact lens wearers (as defined in Section 10.3 Preoperative Procedures)
6. Subjects with diagnosed degenerative visual disorders (e.g., macular degeneration or other retinal disorders) that are predicted to cause visual acuity loss to a level worse than 20/30 Snellen (0.67 decimal) during the study
7. Subjects with conditions associated with increased risk of zonular rupture, including capsular or zonular abnormalities that may lead to IOL decentration or tilt, such as pseudoexfoliation, trauma, or posterior capsule defects
8. Use of systemic or ocular medications that may affect vision, confound the outcome or increase the risk to the subject (e.g., poor dilation or a lack of adequate iris structure to perform standard cataract surgery)
9. Acute, chronic, or uncontrolled systemic or ocular disease or illness that, in the opinion of the investigator, would increase the operative risk or confound the outcome(s) of the study (e.g., immunocompromised, connective tissue disease, suspected glaucoma, glaucomatous changes in the fundus or visual field, ocular inflammation, etc.). Note: controlled ocular hypertension without glaucomatous changes (optic nerve cupping and visual field loss) is acceptable.
10. Planned monovision correction (one eye designated for near correction).
11. Patients who are pregnant or nursing.
12. Severe or unstable systemic disease that may affect the heart, liver, kidney, lung, endocrine (including thyroid insufficiency), blood, or psychoneurological dysfunction
13. Any other systemic or ocular disease that, in the opinion of the investigator, may affect the patient's eligibility for the study, affect visual acuity or may require surgical intervention during the course of the study (e.g., macular degeneration, cystoid macular edema, diabetic retinopathy, etc.).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2021-11-24 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
percentage of eyes that are measured at the 1-week postoperative visit to demonstrate ≤10º change from the intended IOL axis at the end of surgery | 1 week

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Surgical Vision Clinical Trials, Study Director — Johnson & Johnson Surgical Vision
Locations (1):
- The Second Affiliated Hospital Zhejiang University School of Medicine, Hangzhou, China

IPD SHARING:
Plan to Share IPD: Yes
Johnson & Johnson Medical Devices Companies have an agreement with the Yale Open Data Access (YODA) Project to serve as the independent review panel for evaluation of requests for clinical study reports and participant level data from investigators and physicians for scientific research that will advance medical knowledge and public health. Requests for access to the study data can be submitted through the YODA project site at http://yoda.yale.edu
URL: http://yoda.yale.edu